CLINICAL TRIAL: NCT00393939
Title: A Randomized Phase 3 Study Of Docetaxel In Combination With Sunitinib Versus Docetaxel In The First-Line Treatment Of Advanced Breast Cancer Patients
Brief Title: Study Of Sunitinib In Combination With Docetaxel Vs Docetaxel In Patients With Advanced Breast Cancer
Acronym: SUN 1064
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A6181064
Record Dates: First submitted 2006-10-30; First posted 2006-10-31 (Estimated); Results first posted 2011-02-28 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Breast Neoplasms
Keywords: advanced breast cancer; sunitinib; docetaxel; Phase 3
MeSH Terms: conditions — Breast Neoplasms | interventions — Sunitinib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: Sunitinib malate
- B (Active Comparator)
  Interventions: Drug: Taxotere

INTERVENTIONS:
Drug: Sunitinib malate — Sunitinib 37.5 mg daily by oral capsule in schedule 2/1 with Docetaxel 75 mg/m2 every 3 weeks or 37. 5 mg daily in continuous dosing (in absence of docetaxel)
  Arms: A
Drug: Taxotere — Docetaxel 100 mg/m2 every 3 weeks in the comparator arm
  Arms: B

SUMMARY:
This is a phase 3 randomized trial evaluating the anti-tumor activity and safety of sunitinib combined with docetaxel versus docetaxel, administered as first-line treatment, in patients with unresectable locally recurrent or metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer with evidence of unresectable locally recurrent, or metastatic disease
* Her-2 negative tumors

Exclusion Criteria:

* Patients for whom docetaxel is contraindicated
* Clinical presentation of inflammatory carcinoma with no other measurable disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 594 (Actual)
Dates: Start 2007-02; Primary Completion 2010-02 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (128):
- United States (8):
  - Pfizer Investigational Site, Berkely, California
  - Pfizer Investigational Site, Shreveport, Louisiana
  - Pfizer Investigational Site, Beaumont, Texas
  - Pfizer Investigational Site, Burleson, Texas
  - Pfizer Investigational Site, Cleburne, Texas
  - Pfizer Investigational Site, Fort Worth, Texas
  - Pfizer Investigational Site, Mineral Wells, Texas
  - Pfizer Investigational Site, Weatherford, Texas
- Argentina (3):
  - Pfizer Investigational Site, La Plata, Buenos Aires
  - Pfizer Investigational Site, Pergamino, Buenos Aires
  - Pfizer Investigational Site, Burnos Aires
- Australia (7):
  - Pfizer Investigational Site, Tweed Heads, New South Wales
  - Pfizer Investigational Site, Redcliffe, Queensland
  - Pfizer Investigational Site, Adelaide, South Australia
  - Pfizer Investigational Site, Brighton, Victoria
  - Pfizer Investigational Site, Malvern, Victoria
  - Pfizer Investigational Site, Ringwood East, Victoria
  - Pfizer Investigational Site, Perth, Western Australia
- Austria (2):
  - Pfizer Investigational Site, Salzburg
  - Pfizer Investigational Site, Vienna
- Belgium (3):
  - Pfizer Investigational Site, Brasschaat
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Verviers
- Canada (4):
  - Pfizer Investigational Site, Surrey, British Columbia
  - Pfizer Investigational Site, Greater Sudbury, Ontario
  - Pfizer Investigational Site, Hamilton, Ontario
  - Pfizer Investigational Site, Kingston, Ontario
- Colombia (3):
  - Pfizer Investigational Site, Bogota, Cundinamarca
  - Pfizer Investigational Site, Pereira, Risaralda Department
  - Pfizer Investigational Site, Cali, Valle del Cauca Department
- Czechia (3):
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, Nový Jičín
  - Pfizer Investigational Site, Prague
- Finland (2):
  - Pfizer Investigational Site, Tampere
  - Pfizer Investigational Site, Turku
- France (9):
  - Pfizer Investigational Site, Bordeaux
  - Pfizer Investigational Site, Dijon
  - Pfizer Investigational Site, Nantes
  - Pfizer Investigational Site, Reims
  - Pfizer Investigational Site, Saint-Cloud
  - Pfizer Investigational Site, Saint-Priest-en-Jarez
  - Pfizer Investigational Site, Strasbourg
  - Pfizer Investigational Site, Tours
  - Pfizer Investigational Site, Villejuif
- Germany (12):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Chemnitz
  - Pfizer Investigational Site, Essen
  - Pfizer Investigational Site, Hildesheim
  - Pfizer Investigational Site, Karlsruhe
  - Pfizer Investigational Site, Leverkusen
  - Pfizer Investigational Site, Magdeburg
  - Pfizer Investigational Site, Marburg
  - Pfizer Investigational Site, Oldenburg
  - Pfizer Investigational Site, Ravensburg
  - Pfizer Investigational Site, Rosenheim
  - Pfizer Investigational Site, Würzburg
- Hungary (3):
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Kaposvár
  - Pfizer Investigational Site, Szentes
- Ireland (2):
  - Pfizer Investigational Site, Dublin
  - Pfizer Investigational Site, Galway
- Italy (12):
  - Pfizer Investigational Site, Catania
  - Pfizer Investigational Site, Cattolica (RN)
  - Pfizer Investigational Site, Cefalu' (PA)
  - Pfizer Investigational Site, Chieti Scalo
  - Pfizer Investigational Site, Lecce
  - Pfizer Investigational Site, Livorno
  - Pfizer Investigational Site, Macerata
  - Pfizer Investigational Site, Napoli
  - Pfizer Investigational Site, Palermo
  - Pfizer Investigational Site, Pavia
  - Pfizer Investigational Site, Rimini
  - Pfizer Investigational Site, Roma
- Netherlands (3):
  - Pfizer Investigational Site, Nijmegen
  - Pfizer Investigational Site, Utrecht
  - Pfizer Investigational Site, Venlo
- Pfizer Investigational Site, Panama City, Provincia de Panamá, Panama
- Poland (5):
  - Pfizer Investigational Site, Gdansk
  - Pfizer Investigational Site, Lubin
  - Pfizer Investigational Site, Poznan
  - Pfizer Investigational Site, Rybnik
  - Pfizer Investigational Site, Warsaw
- Portugal (4):
  - Pfizer Investigational Site, Coimbra
  - Pfizer Investigational Site, Lisbon
  - Pfizer Investigational Site, Porto
  - Pfizer Investigational Site, Santa Maria da Feira
- Romania (3):
  - Pfizer Investigational Site, Cluj-Napoca, Cluj
  - Pfizer Investigational Site, Craiova, Dolj
  - Pfizer Investigational Site, Bucharest, Sector 2
- Russia (3):
  - Pfizer Investigational Site, Kuzmolovo, Vsevolozhsk District, Leningradskaya Oblast'
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Saint Petersburg
- Slovakia (3):
  - Pfizer Investigational Site, Banská Bystrica
  - Pfizer Investigational Site, Bratislava
  - Pfizer Investigational Site, Nitra
- South Korea (2):
  - Pfizer Investigational Site, Goyang-si, Gyeonggi-do
  - Pfizer Investigational Site, Seoul
- Spain (9):
  - Pfizer Investigational Site, Palma de Mallorca, Balearic Islands
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Santiago de Compostela, La Coruña
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Santa Cruz de Tenerife, Santa Cruz de Tenerife
  - Pfizer Investigational Site, Dos Hermanas, Sevilla
  - Pfizer Investigational Site, Toledo, Toledo
  - Pfizer Investigational Site, Valencia, Valencia
  - Pfizer Investigational Site, Zaragoza, Zaragoza
- Sweden (4):
  - Pfizer Investigational Site, Helsingborg
  - Pfizer Investigational Site, Karlstad
  - Pfizer Investigational Site, Stockholm
  - Pfizer Investigational Site, Uppsala
- Turkey (Türkiye) (3):
  - Pfizer Investigational Site, Ankara
  - Pfizer Investigational Site, Gaziantep
  - Pfizer Investigational Site, Istanbul
- Ukraine (5):
  - Pfizer Investigational Site, Dnipropetrovsk
  - Pfizer Investigational Site, Donetsk
  - Pfizer Investigational Site, Ivano-Frankivsk
  - Pfizer Investigational Site, Kyiv
  - Pfizer Investigational Site, Lviv
- United Kingdom (10):
  - Pfizer Investigational Site, Cheltenham, Gloucestershire
  - Pfizer Investigational Site, Maidstone, Kent
  - Pfizer Investigational Site, Manchester, M20 4bx
  - Pfizer Investigational Site, Metropolitan Borough of Wirral, Merseyside
  - Pfizer Investigational Site, Shrewsbury, Shropshire
  - Pfizer Investigational Site, Telford, Shropshire
  - Pfizer Investigational Site, Guildford, Surrey
  - Pfizer Investigational Site, Worthing, West Sussex
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Wolverhampton

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181064&StudyName=Study%20Of%20Sunitinib%20In%20Combination%20With%20Docetaxel%20Vs%20Docetaxel%20In%20Patients%20With%20Advanced%20Breast%20Cancer

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 594 participants enrolled in study; 1 participant withdrew consent prior to treatment. In accordance with French law, that participant's data was not used in the analyses.
Groups:
- Docetaxel + Sunitinib: Sunitinib 37.5 milligrams (mg) daily by oral capsule for 2 weeks followed by a 1-week off-treatment period (Schedule 2/1) with docetaxel 75 milligrams per square meter (mg/m^2) every 3 weeks, or sunitinib 37.5 mg daily in continuous dosing (in absence of docetaxel), or docetaxel 100 mg/m^2 every 3 weeks (in absence of sunitinib).
- Docetaxel: Docetaxel 100 mg/m^2 every 3 weeks
Period: Overall Study
Arm/Group | Docetaxel + Sunitinib | Docetaxel
Started | 296 | 297
Treated | 295 | 293
Completed | 0 | 0
Not Completed | 296 | 297
Not completed — Protocol Violation | 1 | 1
Not completed — Lost to Follow-up | 2 | 4
Not completed — Death | 10 | 4
Not completed — Sponsor | 5 | 13
Not completed — Objective progression or relapse | 239 | 223
Not completed — Withdrawal by Subject | 2 | 7
Not completed — Other | 37 | 45

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Docetaxel + Sunitinib | Docetaxel | Total
Number analyzed (Participants) | 296 | 297 | 593
Age Continuous [Mean (Standard Deviation); unit: Years] | 54.3 (9.74) | 55.1 (10.36) | 54.7 (10.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 296 | 297 | 593
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS defined as time from date of randomization to date of the first documentation of objective tumor progression or death due to any cause, whichever occurred first. PFS calculated as (Months) = (first event date minus randomization date plus 1) divided by 30.4.
Time Frame: Baseline up to Month 33
Population: Intent-to-Treat (ITT) Population: all randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel + Sunitinib | Docetaxel
Number analyzed (Participants) | 296 | 297
months
  Independent radiology assessment | 8.6 [8.2 to 10.3] | 8.3 [7.7 to 9.6]
  Investigator's assessment | 8.2 [7.3 to 8.6] | 6.9 [6.5 to 7.3]
Statistical Analysis 1: Comparison: Docetaxel + Sunitinib vs Docetaxel; Independent radiology assessment; Test type: Superiority or Other; p = 0.2651, Log Rank — 1-sided stratified log-rank test adjusted for baseline stratification factors (number of metastatic sites, estrogen receptor status, and disease-free interval from prior adjuvant treatment); Hazard Ratio (HR) = 0.9222, 95% CI 2-sided [0.7156 to 1.1885]
Statistical Analysis 2: Comparison: Docetaxel + Sunitinib vs Docetaxel; Investigator's assessment; Test type: Superiority or Other; p = 0.0753, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.8560, 95% CI 2-sided [0.6921 to 1.0589]

2. Secondary Outcome: Percentage of Participants With Objective Response
Description: Percentage of participants with objective response based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). CR defined as the disappearance of all tumor lesions (target and non-target). PR defined as greater than or equal to 30 percent (≥30%) decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions with a non-progressive disease status of the non-target lesions.
Time Frame: Baseline up to Month 33
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Docetaxel + Sunitinib | Docetaxel
Number analyzed (Participants) | 296 | 297
percentage of participants
  Independent radiology assessment | 51.0 | 39.1
  Investigator's assessment | 52.7 | 43.8
Statistical Analysis 1: Comparison: Docetaxel + Sunitinib vs Docetaxel; Independent radiology assessment; Test type: Superiority or Other; p = 0.0018, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.65, 95% CI 2-sided [1.17 to 2.33]
Statistical Analysis 2: Comparison: Docetaxel + Sunitinib vs Docetaxel; Investigator's assessment; Test type: Superiority or Other; p = 0.0172, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.44, 95% CI 2-sided [1.03 to 2.02]

3. Secondary Outcome: Duration of Response (DR)
Description: DR defined as time from first objective documentation of complete or partial response that was subsequently confirmed to first documentation of disease progression or to death due to any cause, whichever occurred first. DR calculated (Months) = (the date of the first documentation of objective tumor progression or death due to any cause minus the date of the first CR or PR that was subsequently confirmed plus 1) divided by 30.4.
Time Frame: Baseline up to Month 33
Population: ITT population. Number of participants analyzed = number of participants with confirmed objective tumor response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel + Sunitinib | Docetaxel
Number analyzed (Participants) | 156 | 130
months
  Independent radiology asssessment (n=151, 116) | 7.5 [6.3 to 9.8] | 7.2 [5.7 to 9.9]
  Investigator's assessment (n=156, 130) | 6.9 [5.8 to 7.1] | 5.8 [5.0 to 7.0]

4. Secondary Outcome: Overall Survival (OS)
Description: Time from randomization to date of death due to any cause. OS calculated as (Months) = (death date minus date of first dose of study medication plus 1) divided by 30.4. For participants who were alive, overall survival was censored at last contact.
Time Frame: Baseline to date of death from any cause (up to Month 33)
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel + Sunitinib | Docetaxel
Number analyzed (Participants) | 296 | 297
months | 26.0 [22.5 to 32.1] | 28.9 [25.5 to 33.4]
Statistical Analysis 1: Comparison: Docetaxel + Sunitinib vs Docetaxel; Test type: Superiority or Other; p = 0.8933, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.1539, 95% CI 2-sided [0.9209 to 1.4458]

5. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionaire-C30 (EORTC- QLQ-C30) Score
Description: EORTC QLQ-C30 measured 5 functional domains (physical, role, cognitive, emotional, and social), global health status, and symptom scales of fatigue, pain, nausea and vomiting, dyspnoea, loss of appetite, insomnia, constipation and diarrhea, and financial difficulties. For functional domains and global health status, scores ranged from 0 to 100 where higher scores represented a better level of functioning. For symptoms scales, scores ranged from 0 to 100 where higher scores represented a greater degree of symptoms. Change from baseline = score for Cycle/Day minus baseline score.
Time Frame: Baseline, every 6 weeks up to end of treatment or early termination (up to Month 33)
Population: ITT population; data not analyzed because study failed its primary endpoint.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Docetaxel + Sunitinib | Docetaxel
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline in EORTC-QLQ Breast Cancer Module (EORTC-QLQ-BR23) Score
Description: EORTC-QLQ-BR23 measured multi-item functional scales for body image, sexual functioning, sexual enjoyment, and future perspective and measured single item symptoms scales which assessed systemic therapy side effects, breast symptoms, arm symptoms, and upset by hair loss. For functional scales, scores ranged from 0 to 100 where higher scores represented a better level of functioning. For symptoms scales, scores ranged from 0 to 100 where higher scores represented a greater degree of symptoms. Change from baseline = score for Cycle/Day minus baseline score.
Time Frame: Baseline, every 6 weeks up to end of treatment or early termination (up to Month 33)
Population: ITT population; data not analyzed because study failed its primary endpoint.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Docetaxel + Sunitinib | Docetaxel
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change From Baseline European Quality of Life 5-dimensional Self-Report Questionnaire (EQ-5D) Score
Description: EQ-5D: standardized, participant-administered 2 part measure of health outcome. Part 1: descriptive profile for 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), used 3 levels (no, some, extreme problems) and a single index value characterized current health status using formula that weighted the dimensions. Part 2: overall rating of participant's current health used Visual Analog Scale with endpoints labeled 'best imaginable health state' and 'worst imaginable health state'. Change from baseline = score for Cycle/Day minus baseline score.
Time Frame: Baseline, every 6 weeks up to end of treatment or early termination (up to Month 33)
Population: ITT population; data not analyzed because study failed its primary endpoint.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Docetaxel + Sunitinib | Docetaxel
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Docetaxel + Sunitinib | Docetaxel
Serious Adverse Events (participants affected / at risk) | 112/295 | 79/293
Other Adverse Events (participants affected / at risk) | 290/295 | 291/293
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel + Sunitinib (N=295) | Docetaxel (N=293)
Anaemia (Blood and lymphatic system disorders) | 4 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 20 | 13
Leukopenia (Blood and lymphatic system disorders) | 5 | 7
Lymphatic disorder (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 11 | 16
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrioventricular block (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac disorder (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1
Conjunctivitis (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 1
Cheilitis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 2
Diverticular perforation (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 6
Oesophagitis ulcerative (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Periproctitis (Gastrointestinal disorders) | 2 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 3 | 2
Vomiting (Gastrointestinal disorders) | 4 | 4
Adverse drug reaction (General disorders) | 1 | 0
Asthenia (General disorders) | 4 | 1
Chest pain (General disorders) | 1 | 0
Death (General disorders) | 1 | 0
Disease progression (General disorders) | 6 | 4
Fatigue (General disorders) | 2 | 1
General physical health deterioration (General disorders) | 5 | 4
Impaired healing (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 2 | 1
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 0 | 2
Pyrexia (General disorders) | 10 | 5
Cholestasis (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1
Catheter site infection (Infections and infestations) | 2 | 1
Cellulitis (Infections and infestations) | 1 | 0
Clostridial infection (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 3
Diverticulitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Groin infection (Infections and infestations) | 1 | 0
Haematoma infection (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 2 | 3
Localised infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Necrotising fasciitis (Infections and infestations) | 1 | 0
Neutropenic infection (Infections and infestations) | 3 | 3
Neutropenic sepsis (Infections and infestations) | 3 | 3
Osteomyelitis (Infections and infestations) | 1 | 0
Peridiverticular abscess (Infections and infestations) | 0 | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 5
Pneumonia primary atypical (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Rectal abscess (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 2 | 1
Sinusitis (Infections and infestations) | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 2 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Blood culture positive (Investigations) | 0 | 1
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bone disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Endometrial sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Psychomotor skills impaired (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Tremor (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 4 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 2 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 2 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1
Embolism (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 4 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 1 | 0
Device dislocation (General disorders) | 1 | 0
Device related infection (Infections and infestations) | 2 | 0
Paronychia (Infections and infestations) | 0 | 1
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel + Sunitinib (N=295) | Docetaxel (N=293)
Anaemia (Blood and lymphatic system disorders) | 67 | 50
Leukopenia (Blood and lymphatic system disorders) | 77 | 83
Neutropenia (Blood and lymphatic system disorders) | 165 | 144
Thrombocytopenia (Blood and lymphatic system disorders) | 45 | 5
Tachycardia (Cardiac disorders) | 21 | 12
Hypothyroidism (Endocrine disorders) | 17 | 2
Conjunctivitis (Eye disorders) | 20 | 16
Eyelid oedema (Eye disorders) | 16 | 2
Lacrimation increased (Eye disorders) | 69 | 50
Abdominal pain (Gastrointestinal disorders) | 36 | 25
Abdominal pain upper (Gastrointestinal disorders) | 22 | 14
Constipation (Gastrointestinal disorders) | 57 | 51
Diarrhoea (Gastrointestinal disorders) | 177 | 111
Dry mouth (Gastrointestinal disorders) | 33 | 19
Dyspepsia (Gastrointestinal disorders) | 70 | 24
Gastritis (Gastrointestinal disorders) | 18 | 10
Gingivitis (Gastrointestinal disorders) | 16 | 2
Nausea (Gastrointestinal disorders) | 119 | 114
Stomatitis (Gastrointestinal disorders) | 96 | 75
Vomiting (Gastrointestinal disorders) | 59 | 65
Asthenia (General disorders) | 99 | 88
Face oedema (General disorders) | 37 | 12
Fatigue (General disorders) | 127 | 101
Mucosal inflammation (General disorders) | 82 | 59
Oedema (General disorders) | 32 | 16
Oedema peripheral (General disorders) | 67 | 93
Pyrexia (General disorders) | 56 | 48
Infection (Infections and infestations) | 16 | 9
Nasopharyngitis (Infections and infestations) | 28 | 18
Alanine aminotransferase increased (Investigations) | 21 | 10
Aspartate aminotransferase increased (Investigations) | 20 | 10
Haemoglobin decreased (Investigations) | 18 | 7
Weight decreased (Investigations) | 21 | 13
Decreased appetite (Metabolism and nutrition disorders) | 94 | 71
Hyperglycaemia (Metabolism and nutrition disorders) | 13 | 20
Arthralgia (Musculoskeletal and connective tissue disorders) | 45 | 65
Back pain (Musculoskeletal and connective tissue disorders) | 27 | 31
Bone pain (Musculoskeletal and connective tissue disorders) | 35 | 38
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 26 | 29
Myalgia (Musculoskeletal and connective tissue disorders) | 53 | 72
Pain in extremity (Musculoskeletal and connective tissue disorders) | 40 | 36
Dizziness (Nervous system disorders) | 18 | 15
Dysgeusia (Nervous system disorders) | 89 | 68
Headache (Nervous system disorders) | 48 | 38
Neuropathy peripheral (Nervous system disorders) | 41 | 50
Paraesthesia (Nervous system disorders) | 22 | 27
Peripheral sensory neuropathy (Nervous system disorders) | 46 | 54
Insomnia (Psychiatric disorders) | 29 | 24
Cough (Respiratory, thoracic and mediastinal disorders) | 45 | 27
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 63 | 54
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 71 | 16
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 22 | 10
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 20 | 16
Alopecia (Skin and subcutaneous tissue disorders) | 178 | 188
Dry skin (Skin and subcutaneous tissue disorders) | 28 | 15
Erythema (Skin and subcutaneous tissue disorders) | 28 | 18
Nail disorder (Skin and subcutaneous tissue disorders) | 44 | 61
Onycholysis (Skin and subcutaneous tissue disorders) | 6 | 17
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 124 | 26
Pruritus (Skin and subcutaneous tissue disorders) | 17 | 31
Rash (Skin and subcutaneous tissue disorders) | 49 | 50
Flushing (Vascular disorders) | 14 | 18
Hypertension (Vascular disorders) | 36 | 3
Lymphoedema (Vascular disorders) | 14 | 19
Febrile neutropenia (Blood and lymphatic system disorders) | 29 | 22
Chest pain (General disorders) | 15 | 11
Pain (General disorders) | 15 | 12
Cystitis (Infections and infestations) | 6 | 16
Skin toxicity (Skin and subcutaneous tissue disorders) | 15 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.